CLINICAL TRIAL: NCT01289509
Title: A Randomized, Open-Label, 4-Way Crossover Replicate Design Study to Evaluate the Relative Bioavailability and Intra-Subject Variability of Two Lots of E5501 40 mg Tablets Administered Twice as Single Oral Doses to Healthy Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Intra-Subject Variability of Two Lots of E5501 40 mg Tablets Administered Twice as Single Oral Doses to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E5501-A001-007
Record Dates: First submitted 2011-01-27; First posted 2011-02-03 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Idiopathic Thrombocytopenia Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

ARMS (2):
- Experimental 1 (Experimental): Drug: E5501
  Interventions: Drug: E5501
- Experimental 2 (Experimental): Drug: E5501
  Interventions: Drug: Drug: E5501

INTERVENTIONS:
Drug: E5501 — Lot P01010ZZA (test) single oral doses of 40 mg tablets.
  Arms: Experimental 1
Drug: Drug: E5501 — Lot P97001ZZB (reference) single oral doses of 40 mg tablets.
  Arms: Experimental 2

SUMMARY:
The purpose of this study is to evaluate the relative bioavailability (BA) of two lots of E5501 40 mg tablets administered twice as single oral doses to healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, open label, 4- way crossover, replicate design study to evaluate the bioavailability (BA) of E5501 new Phase 3 formulation Lot P97001ZZB 40 mg tablet manufactured July, 2009 (Treatment A ,reference drug) relative to Lot P01010ZZA 40 mg tablet manufactured January, 2010 (Treatment B, test drug) administered to 42 healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy adult male or female subjects age greater than or equal to 18 years and less than or equal to 55 years old.
* Body mass index greater than or equal to 18 kg/m2 and less than or equal to 32 kg/m2 at the time of screening.
* Platelet count between 120x109/L and 250x109/L.
* Women of childbearing potential must agree to use a double barrier method of contraception during the Randomization Phase of the study.

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact the pharmacokinetics (PK)of the study drug.
* Agents associated with thrombotic events (including oral contraceptives) must be discontinued within 30 days of the first study drug administration.
* Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history, e.g., history of splenectomy.
* History of venous or arterial thrombotic disease or other hypercoaguable state.
* Hemoglobin level less than 11.5 g/dL for females and 13.5g /dL for males

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-12; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
• To evaluate the bioavailability (BA) , as measured by AUC point estimates of E5501 40 mg tablet Lot P01010ZZA (test) relative to E5501 40 mg tablet Lot P97001ZZB (reference). | 96 hours post-dose
To evaluate the bioavailability, as measured by Cmax point estimates of E5501 40 mg tablet Lot P01010ZZA (test) relative to E5501 40 mg tablet Lot P97001ZZB (reference). | 96 hours post dose

SECONDARY OUTCOMES:
• To assess the intra-subject and inter-subject variability in Cmax following replicate dosing with E5501 40 mg lots | 10 weeks
• To assess the intra-subject and inter-subject variability in AUC(0-inf) following replicate dosing with E5501 40 mg lots. | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Johnson, Study Director — Eisai Inc.
Locations (1):
- PRA, Lenexa, Kansas, United States